CLINICAL TRIAL: NCT05188846
Title: Caries Arresting Treatment Using Silver Diamine Fluoride (SDF) Versus SDF Modified Atraumatic Restorative Technique (SMART) for Management of Carious Vital Primary Teeth: A Randomized Clinical Trial
Brief Title: Caries Arresting in Primary Molar Teeth Using SDF VS ART
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ola Adel Abdelfadil Ahmed (Other)
Responsible Party: Sponsor-Investigator, Ola Adel Abdelfadil Ahmed, master student, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDF VS ART
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDF (Experimental)
  Interventions: Other: SDF
- SDF + ART ( SMART technique ) (Active Comparator)
  Interventions: Other: SDF + ART (SMART technique )

INTERVENTIONS:
Other: SDF — 1. Group 1: cleaning the occlusal surface to be treated with toothbrush. Decayed tissue from the affected teeth will not be removed for the SDF group.
  Clinical procedure for SDF application: it will apply according to the SDF manufacturer Instructions as follows:(1) the surrounding gingival tissues and lips will be protected with petroleum jelly to avoid staining and irritation,(2) the affected tooth will be isolated and keep dry with cotton rolls and saliva ejectors, (3) one drop of SDF (SDI RIVA STAR ), will be placed into a disposable dish, (4) SDF will be applied with a micro-sponge directly to the affected tooth surface(s), (5) allowed to soak in for 2 min, then air-dried. Then will be followed by the Potassium iodide (KI) liquid to decrease discoloration caused by SDF. The KI liquid will be reapplied until no more white perception observed to form.
  Arms: SDF
Other: SDF + ART (SMART technique ) — 2. Group 2: SDF+ART clinical procedure: (1)cleaning the occlusal surface to be treated with toothbrush.,(2) carious dentin will be removed using a small excavator (Spoon excavator ),(3) the cavity will be cleaned and dried, (4)cavity walls and floor will be conditioned for 10s, then washed and dried, (5) SDF will be applied as mentioned above followed by cavity restoration using resin-reinforced glass ionomer restorative material (SDI RIVA ).
  Arms: SDF + ART ( SMART technique )

SUMMARY:
This study aimed to evaluate the oral health related quality of life ( OHRQoL), during caries management in children with vital carious primary teeth with no signs of irreversible pulpitis using SDF alone or SDF in combination with ART, using Early Childhood Oral Health Impact Scale (ECOHIS).

DETAILED DESCRIPTION:
Early childhood caries (ECC) is a type of dental caries in the teeth of infants and children that is represented as one of the most prevalent dental problems in this period, which can lead to pain, infection, interference with eating.

According to the ADA, (ECC) is described as "the presence of one or more decayed ( cavitated or non cavitated lesions), missing (due to caries), or filled tooth surfaces in any primary tooth" in children.

Overall, 50% of children have one or more decayed primary teeth by the end of toddler age, but the importance of these teeth should not be neglected, because, healthy teeth in childhood have an important role in the eruption of healthy permanent teeth, healthy nutrition, and aesthetic appearance.

Conventional treatment methods (drill and fill) involve the use of rotary burs under local anesthesia which develops pain and needs cooperative child and highly trained dental health personnel and consider an invasive technique, on the other hand (ART) is an approach to increase accessibility to restorative treatment, inexpensive and can be employed in regions without electricity and running water. In addition, ART is a minimally invasive treatment that requires no rotary instruments or local anesthesia to remove decayed tissue before sealing the cavity with high viscosity glass ionomer cement (GIC).

(SDF), a low-cost cariostatic agent and a noninvasive method for caries management, treatment with SDF are easy, effective, and well accepted, it is also an alternative to traditional restorative treatment and may influence the reduction of untreated carious lesions in childhood

ELIGIBILITY:
Inclusion Criteria: • Age: 4-6 years old age.

* Both genders.
* Decayed vital primary molars (asymptomatic teeth with active single-surface lesions, vital pulp no signs of irreversible pulpitis) .

Exclusion Criteria:

* History of systemic conditions.
* Allergy to silver.
* Oral ulceration.
* Teeth with proximal or multi-surfaces caries, pulp pathology.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2022-01-25 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
ECOHIS | 6 month
  Early Childhood Oral Health Impact Scale.

SECONDARY OUTCOMES:
- Clinical effectiveness Caries arrestment/ treatment | 6 month
  International Caries Detection and Assessment System (ICDAS II)

CONTACTS AND LOCATIONS:
Overall Officials: Nevine Waly, Professor, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: No